CLINICAL TRIAL: NCT05912907
Title: Potassium Nitrate in Polycarboxylate Versus Mineral Trioxide Aggregate as a Direct Pulp Capping in Young Permanent Molars
Brief Title: Potassium Nitrate in Polycarboxylate as a Direct Pulp Capping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 532
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases | interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- potassium nitrate in polycarboxilate cement (Experimental)
  Interventions: Other: potassium nitrate in polycarboxilate cement
- Mineral Trioxide Aggregate (Active Comparator)
  Interventions: Other: potassium nitrate in polycarboxilate cement

INTERVENTIONS:
Other: potassium nitrate in polycarboxilate cement — 5% potassium nitrate in polycarboxylate; pre-weighed 95 mg zinc oxide powder and 5mg of KNO3 will be placed on a glass slab followed by mixing by polyacrylic acid (liquid) in a 1:1 P/L ratio

SUMMARY:
The study aimed to compare potassium nitrate in polycarboxylate cement to mineral trioxide aggregate as a direct pulp capping material of young permanent teeth in patients from 7 to 10 ears

ELIGIBILITY:
Inclusion Criteria:

* 7-10 years of children
* Healthy children classified as ASA I or II
* Asymptomatic vital immature mandibular first molar with extensive and deep caries
* Signs and symptoms of reversible pulpitis

Exclusion Criteria:

* Necrotic teeth or teeth with irreversible pulpitis
* Medically compromised children

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
clinical success rate | 24 months
  Absence of pain, sensitivity to percussion, fistula or sinus tract, mobility
Radiographic success rate | 24 months
  Absence of periapical radiolucency, internal root resorption, external root resorption

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Al Minyā, Egypt